CLINICAL TRIAL: NCT04977739
Title: Research on the Application and Mechanism of New Biological Probes in Biomedicine
Status: Completed | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2021-007
Record Dates: First submitted 2021-07-14; First posted 2021-07-27 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2021-06

CONDITIONS: Tumors; Cardiovascular Diseases; Respiratory System Diseases; Digestive System Diseases; Endocrine System Diseases; Metabolic Diseases; Immune System Diseases; Urinary System Diseases; Nervous System Diseases; Blood Diseases; Infectious Diseases
MeSH Terms: conditions — Neoplasms; Cardiovascular Diseases; Respiratory Tract Diseases; Digestive System Diseases; Endocrine System Diseases; Metabolic Diseases; Immune System Diseases; Urologic Diseases; Nervous System Diseases; Hematologic Diseases; Communicable Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- those with a condition
  Interventions: Diagnostic Test: No intervention
- those without a condition
  Interventions: Diagnostic Test: No intervention

INTERVENTIONS:
Diagnostic Test: No intervention — No intervention

SUMMARY:
Fluorescence is one of the most commonly used research and detection techniques in the field of biomedical science. The characteristics of fluorescent probe directly affect the performance and application of fluorescence analysis and imaging. Aggregation-Caused Quenching has limited the application of traditional fluorescent probes to some extent. This project intends to systematically evaluate the detection efficiency of new methods through the detection of biomarkers in clinical samples and the comparison with the detection methods of traditional biomarkers, so as to provide theoretical and experimental basis for the establishment of fast and simple biomarker detection technologies with new biological probes.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form voluntarily.
* Age 18-70 years old.
* High expression (positive) group: The results of multiple laboratory tests indicate that the marker is higher than the normal range.
* Low expression (negative) healthy volunteer group: those with no underlying diseases and no abnormalities in the physical examination.
* Have routine examination to check the remaining body fluid samples, and the body fluid samples are not contaminated.

Exclusion Criteria:

* Accompanied by other inflammations.
* The data of the subject is not complete, or the collection of cases is incomplete due to other reasons.
* The researcher judged that it was not suitable to participate in this research.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: NanFang Hospital samples
Sampling Method: Probability Sample
Enrollment: 737 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
signal intensity of the probes | one day

CONTACTS AND LOCATIONS:
Overall Officials: Bo Situ, Study Director — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China